CLINICAL TRIAL: NCT06789887
Title: Increasing Access to Evidenced-Based PTSD Treatment in the Military: Behavioral Health Technician Delivered Written Exposure Therapy
Brief Title: Behavioral Health Technician Delivered Written Exposure Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); Brooke Army Medical Center (U.S. Federal Agency); Naval Hospital Camp Pendleton (U.S. Federal Agency); NDRI-USA, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCA0011
Record Dates: First submitted 2025-01-06; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Post Traumatic Stress Disorder; Written Exposure Therapy
Keywords: PTSD; Post Traumatic Stress Disorder; Behavioral Health Technician; Written Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (Active Comparator): Participants in this arm will receive usually prescribed behavioral health treatment.
  Interventions: Behavioral: Treatment as Usual (TAU)
- Treatment As Usual (TAU) and Written Exposure Therapy (WET) (Experimental): Participants in this arm will receive the usually prescribed behavioral health treatment as well as 5 total sessions of Written Exposure Therapy with a Behavioral Health Technician.
  Interventions: Behavioral: Written Exposure Therapy; Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Written Exposure Therapy (WET) is a 5-session, trauma-focused intervention in which individuals write about their traumatic experience following scripted instructions.
  Arms: Treatment As Usual (TAU) and Written Exposure Therapy (WET)
Behavioral: Treatment as Usual (TAU) — Treatment as usual (TAU) will be available to all patient participants. Treatment as usual may include various forms of psychotherapy and or medication management.

SUMMARY:
This study has two main goals. First, it aims to test a treatment called written exposure therapy to see if it can help military service members who have posttraumatic stress disorder (PTSD). Second, it aims to test a new way of making this therapy more accessible in military clinics by utilizing task-sharing with Behavioral Health Technicians (BHTs). PTSD is a common and serious issue among service members. Written exposure therapy (WET) has been proven to be effective for improving PTSD that requires five therapy sessions delivered weekly. This study aims to determine:

1. How well does written exposure therapy help to reduce symptoms of posttraumatic stress for service members with PTSD?
2. Is sharing the therapy tasks with behavioral health technicians is a helpful approach for managing behavioral health clinic patient volume and improving patient outcomes?

We plan to recruit a total of 40-59 staff participants, as well as 150 active-duty patient participants with PTSD. We will randomize patient participants to one of two treatment conditions: 1) treatment-as-usual (TAU) or 2) TAU and 5 sessions of WET. Staff and participants will be recruited from two military treatment facilities: 1) Fort Sam Houston in San Antonio (Brooke Army Medical Center) and 2) Camp Pendleton (Naval Hospital at Camp Pendleton).

Consented patient participants will:

* Complete a PTSD interview via telehealth with a study team member to determine if you are eligible for the study
* Be randomly assigned to one of the following conditions: 1) TAU + WET or 2) TAU
* Complete up to 8 weeks of behavioral health treatment (either TAU + WET or TAU)
* Complete self-report measures before, during, and after treatment, and at a 3- and 6-month follow up assessment after the treatment period
* Complete a posttreatment PTSD interview via telehealth with a study team member
* A subset of participants will be asked to complete a brief treatment experience interview posttreatment

Consented staff participants will:

* Participate in an interview about your perceptions of and experiences supporting BHT-delivered WET with a study team member at the VAPAHCS
* A subset of participants will also be asked to participate in a brief staff feedback interview approximately 6 months after their first interview

ELIGIBILITY:
Inclusion Criteria:

Patient participants:

1. Adult active duty personnel ages ≥18
2. Clinically significant PTSD symptoms (CAPS-5 ≥ 25).

Clinic staff participants: Individuals working as BHTs, clinic providers, and clinic leaders working at the behavioral health clinics participating in the study

Exclusion Criteria:

Patient participants:

1. Current suicide or homicide risk meriting crisis intervention
2. Serious mental health symptoms, such as mania, psychosis, alcohol or substance use disorders warranting immediate attention
3. Inability to comprehend the baseline screening questionnaires
4. Definite plans to leave the military within 10 weeks

Clinic staff participants:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS-5) | Change from baseline to immediately post treatment
  The CAPS-5 is a 30-item structured clinical interview that assesses the presence and severity of 20 PTSD symptoms as defined by the DSM-5. It also assess the impact of these symptoms on daily functioning and will be used to evaluate if there is a response to the experimental treatment in this study.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist (PCL-5) | Change from baseline through 6 months post treatment
  The PCL-5 is a 20-item self-report questionnaire designed to assess PTSD symptoms as defined by the DSM-5. This questionnaire will be used to monitor changes before and after treatment, as well as screening patients for PTSD.
Insomnia Severity Index (ISI) | Change from baseline through 6 months post treatment
  The ISI is a seven-item questionnaire that is designed as a screening tool to assess the severity of a patient's insomnia using a Likert-type scale.
Generalized Anxiety Disorder 7-Item (GAD-7) Scale | Change from baseline through 6 months post treatment
  The GAD-7 is a 7-item self-report measure of the severity from mild to severe of symptoms related to generalized anxiety; items correspond to the diagnostic criteria for generalized anxiety disorder.
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline through 6 months post treatment
  The PHQ-9 is a 9-item questionnaire that assesses the severity of affective and somatic symptoms related to depression; items correspond to the diagnostic criteria for major depression disorder.
Life Events Checklist for DSM-5 (LEC-5) | Baseline
  The LEC-5 includes a list of 16 different potentially traumatic life events that that are commonly associated with PTSD symptoms and was designed to facilitate the diagnosis of PTSD. Therefore, it is used as a self-report measure designed to screen for potentially traumatic events in a respondent's lifetime and is typically administered before the CAP-5.
Depressive Symptoms Index-Suicidality Subscale (DSI-SS). | Change from baseline through 6 months post treatment
  The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide.
  Scores on each item range from 0 to 3, with higher scores reflecting greater severity of suicidal ideation.
History of Head Injuries | Baseline
  The History of Head Injuries form is a 3-item screening questionnaire that assesses a participant's history of a head injuries and altered consciousness to determine the worst head injury sustained while deployed. The form captures the total number of injuries during and outside of deployment.
Brief Inventory of Psychosocial Functioning (B-IPF). | Changes from baseline through 6 months post treatment
  The B-IPF is a 7-item measure of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. The B-IPF is an abridged version of the 80-item Inventory of Psychosocial Functioning, a survey that assesses psychosocial functioning but that would be too time-intensive to administer.
Credibility/Expectancy Questionnaire (CEQ) | Immediately after the first treatment session, and immediately after the final treatment session
  The CEQ is a 6-item measure that was designed to assess treatment expectancy and rationale credibility for use of an experimental treatment in clinical outcomes studies.
Net Prompter Score | Post treatment (~6 months post baseline)
  The Net Prompter Score is a single item measures of treatment acceptability that asks respondents to rate the likelihood that they would recommend the efficient treatment to a friend or colleague on a scale from 0-10.
Patient Satisfaction Survey | Post treatment (~6 months post baseline)
  The Patient Satisfaction Survey is an adapted version of the Therapeutic Alliance and Patient Satisfaction survey. For this study, adaptations were made in order to assess satisfaction with the care received by the BHT (5 items; among patient participants assigned to WET + TAU) and providers separately (5 items; among all patient participants).
Treatment Engagement | Through study completion, an average of 2 years
  Treatment engagement will be assessed by the BHTs' supervisor at the clinic who will review administrative data to determine the number of behavioral health appointments completed by each enrolled patient participant. Engagement in TAU for patient participant who receive care in the network will be assessed at posttreatment via participant self-report.
WET Adoption | Through study completion, an average of 2 years
  Adoption will be assessed by examining the proportion of available BHTs who participate in the WET training and who deliver WET to study participants.
WET Fidelity | Through study completion, an average of 2 years
  To assess fidelity to the WET protocol, BHTs will audio record treatment sessions and submit a copy of the written trauma narratives. A random subset of 20% of the WET sessions will be reviewed rated for fidelity. Sessions will be rated using the WET Therapist Adherence and Competence Protocol. Clinicians are rated (yes/no) whether each session task was completed (e.g., "Therapist presented the treatment rationale for writing about traumatic event," "Therapist checked in with participant after writing and inquired how writing session went") and how well the therapist delivered each task (1 = poor to 7 = excellent). An overall competence score is also provided for each session.
Demographics and Military Service Characteristics Form | Baseline.
  This form will be administered to participants to measure standard demographics (race, gender, age) and military service information (e.g., deployment history, rank).